CLINICAL TRIAL: NCT06236659
Title: The Dose-response of Vitamin C-enriched Collagen on Markers of Collagen Synthesis in Middle-Aged Men and Women Following Resistance Exercise
Brief Title: Acute Resistance Exercise and Hydrolyzed Collagen Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rob Erskine (Other)
Collaborators: University of East Anglia (Other)
Responsible Party: Sponsor-Investigator, Rob Erskine, Principal Investigator, Liverpool John Moores University
Organization: Liverpool John Moores University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 19/SPS/049
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Diet; Food; Nutrition
Keywords: Hydrolyzed collagen; Resistance Exercise; Collagen Synthesis; Proline; Glycine

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized cross-over design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Before commencing each experimental intervention, a laboratory technician (independent to the study) made up the three doses of hydrolyzed collagen (HC) and randomly assigned the order of HC dose (Excel 2016, Microsoft, Washington, USA) for each participant. Also, for each intervention, the technician recorded the date, randomly allocated trial number (1, 2 or 3) and corresponding HC dose to blind the investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention for middle-aged men: Consumption of hydrolyzed collagen (HC) with resistance exercise (Experimental): Middle-aged male participants consumed one of three different HC doses (0 grams, 15 grams, or 30 grams) with 4 sets of 10 repetitions of leg press exercise at 10-repetition maximum load in a random order and a seven-day wash-out period interspersed between each trial.
  Interventions: Dietary Supplement: Consumption of three different doses of hydrolyzed collagen (HC) with resistance exercise
- Intervention for middle-aged women: Consumption of hydrolyzed collagen (HC) with resistance exercise (Experimental): The intervention procedure is exactly same as Arm 1 except for the number of visits and doses of HC. Middle-aged female participants were asked to visit the laboratory on the day of highest oestrogen (i.e. ovulation) and provided with 0 g or 30 g HC. Dates for the trials were determined based on self-report of onset of menses and previous menstrual cycle length.
  Interventions: Dietary Supplement: Consumption of two different doses of hydrolyzed collagen (HC) with reistance exercise

INTERVENTIONS:
Dietary Supplement: Consumption of three different doses of hydrolyzed collagen (HC) with resistance exercise — Each intervention lasts for seven hours and while participants consumed HC, performed resistance exercise and rested, 10 x 5 mL blood samples were collected from a superficial forearm vein using a cannula.
  All interventions were performed at the same time of day (08:00 - 15:00).
  Different doses of HC (0 grams, 15 grams and 30 grams) and 50 milligrams vitamin C were dissolved with 250 milliliter water in an opaque bottle. To match calories of 30 grams HC, 34.1 grams and 15.4 grams maltodextrin was used in 0 grams HC and 15 grams HC respectively. Also to mask any potential difference in HC doses, 4 grams non-caloric sweetener was used in all HC doses.
  The details of dietary supplements used are as follows:
  Hydrolysed collagen (Myprotein, Cheshire, UK), Vitamin C powder (Holland and Barrett Retail Limited, Warwickshire, UK), Maltodextrin (Myprotein, Cheshire, UK), and Non-caloric sweetener (Truvia®, SilverSpoon, London, UK)
  Other Names: Resistance exercise and collagen dose-response for middle-aged male participants
  Arms: Intervention for middle-aged men: Consumption of hydrolyzed collagen (HC) with resistance exercise
Dietary Supplement: Consumption of two different doses of hydrolyzed collagen (HC) with reistance exercise — Each intervention lasts for seven hours and while participants consumed HC, performed resistance exercise and rested, 10 x 5 mL blood samples were collected from a superficial forearm vein using a cannula.
  All interventions were performed at the same time of day (08:00 - 15:00).
  Different doses of HC (0 grams, and 30 grams) and 50 milligrams vitamin C were dissolved with 250 milliliter water in an opaque bottle. To match calories of 30 grams HC, 34.1 grams and 15.4 grams maltodextrin was used in 0 grams HC and 15 grams HC respectively. Also to mask any potential difference in HC doses, 4 grams non-caloric sweetener was used in all HC doses.
  The details of dietary supplements used are as follows:
  Hydrolysed collagen (Myprotein, Cheshire, UK), Vitamin C powder (Holland and Barrett Retail Limited, Warwickshire, UK), Maltodextrin (Myprotein, Cheshire, UK), and Non-caloric sweetener (Truvia®, SilverSpoon, London, UK)
  Other Names: Resistance exercise and collagen dose-response for middle-aged female participants
  Arms: Intervention for middle-aged women: Consumption of hydrolyzed collagen (HC) with resistance exercise

SUMMARY:
This study aimed to investigate the effect of different doses of hydrolyzed collagen (HC) with resistance exercise (RE) on whole body collagen synthesis in middle-aged males and females.

DETAILED DESCRIPTION:
This study aimed to investigate the effect of different doses of hydrolyzed collagen (HC) with resistance exercise (RE) on whole body collagen synthesis in healthy middle-aged males and females.

Healthy middle-aged males and females ingested 0 grams, 15 grams or 30 grams HC with 50 milligrams vitamin C 1h prior to performing four sets' leg press RE at 10-repetition maximum load, after which they rested for six hours. Blood samples were collected throughout each trial to analyse procollagen type Ⅰ N-terminal propeptide (PⅠNP, a biomarker of collagen synthesis) and β-isomerized C-terminal telopeptide of type I collagen (β-CTX, a biomarker of collagen breakdown) concentration, and the concentration of 18 amino acids that constitute collagen.

This is the first study to investigate the combined effect of different doses HC with high-intensity RE on whole body collagen synthesis in middle-aged men and women. If 30 grams HC intake with RE does augment collagen synthesis more than RE alone, this suggests that long-term HC intake with chronic RE would be beneficial for tendon health, because collagen is the most abundant protein in tendon.

ELIGIBILITY:
Inclusion Criteria:

* At least 12 months experienced in resistance exercise (including weekly lower body exercise)
* Free from musculoskeletal injury

Exclusion Criteria:

* Having a history of patellar tendon pathology
* Vegan
* Consumed nutritional supplements or medication purported to have beneficial effects on muscle-tendon properties (e.g. antioxidants, protein, etc.)
* Had a sustained a lower limb injury in the previous six months
* Smoker/vaper
* Having reached menopause (only for middle-aged female participants)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change in a marker of collagen synthesis | At rest immediately prior to HC ingestion, 0.5-hour post RE, 1-hour post RE, 2-hour post RE, 4-hour post RE and 6-hour post RE
  Serum procollagen type Ⅰ N-terminal propeptide (PⅠNP) concentrations were measured following 0 grams, 15 grams or 30 grams hydrolyzed collagen (HC) intake with resistance exercise (RE) during all interventions.
Change in a marker of collagen breakdown | At rest, immediately prior to HC ingestion, 0.5-hour post RE, 2-hour post RE and 6-hour post RE
  Plasma β-isomerized C-terminal telopeptide of type I collagen (β-CTX) concentrations were measured following 0 grams, 15 grams or 30 grams hydrolyzed collagen (HC) intake with resistance exercise (RE) during all interventions.

SECONDARY OUTCOMES:
Estrogen concentrations in women in each trial | At rest immediately prior to HC ingestion
  Concentrations of estrogen (17β-estradiol) was measured in each intervention.
Changes in amino acids concentrations in blood | At rest immediately prior to HC ingestion, 0.5-hour post HC ingestion, 1-hour post HC ingestion, 0.5-hour post RE, 1-hour post RE, 2-hour post RE, 4-hour post RE and 6-hour post RE
  Concentration of serum amino acids that constitute collagen was measured following 0 grams, 15 grams or 30 grams hydrolyzed collagen (HC) intake with resistance exercise (RE) during all interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Erskine, Principal Investigator — Liverpool John Moores University
Locations (1):
- Dr Rob Erskine, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT06236659/Prot_SAP_ICF_000.pdf